CLINICAL TRIAL: NCT02404714
Title: A Multi-Center Study of A New Method of Sweat Testing: The CF Quantum® Sweat Test
Brief Title: A Multi-Center Study of the CF Quantum® Sweat Test System
Status: Terminated | Type: Observational
Why Stopped: Study funding has been withdrawn. No adverse safety issues.
Sponsor: Polychrome Medical, Inc. (Industry)
Responsible Party: Sponsor
Other Study IDs: CFQuantum003
Record Dates: First submitted 2015-03-16; First posted 2015-03-31 (Estimated); Last update posted 2018-08-31 (Actual); Status verified 2018-08

CONDITIONS: Cystic Fibrosis
MeSH Terms: conditions — Cystic Fibrosis

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Cross-Sectional
Biospecimen Retention: Samples Without DNA — Sweat samples will be collected per standard sweat testing procedure.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | Unapproved Device: Yes

GROUPS / COHORTS (2):
- CF/CRMS: Subject's with a previous cystic fibrosis or cystic fibrosis related metabolic syndrome (CRMS) diagnosis will receive the institution's standard iontophoresis sweat testing (Gibson-Cooke or Wescor Macroduct) to provide a diagnosis.
  The patient will also receive a sweat test provided by the new CF Quantum Sweat Test System which includes the same process and principal of operation of iontophoretic stimulation, collection and analysis of sweat compared to the standard. The results of the new sweat test and the standard sweat test will be compared. The new sweat test will not be used to diagnose, treat or mitigate the patient's condition. Results are used only to compare to the standard of care.
  Interventions: Device: Iontophoresis sweat test
- NON CF/CRMS: Subject's without a previous cystic fibrosis or cystic fibrosis related metabolic syndrome (CRMS) diagnosis but referred to the sweat test lab on a clinical observation basis by a physician will receive standard iontophoresis sweat testing (Gibson-Cooke or Wescor Macroduct) to provide a diagnosis.
  The patient will also receive a sweat test provided by the new CF Quantum Sweat Test System which includes the same process and principal of operation of iontophoretic stimulation, collection and analysis of sweat compared to the standard. The results of the new sweat test and the standard sweat test will be compared. The new sweat test will not be used to diagnose, treat or mitigate the patient's condition. Results are used only to compare to the standard of care.
  Interventions: Device: Iontophoresis sweat test

INTERVENTIONS:
Device: Iontophoresis sweat test — The intervention is iontophoretic sweat testing which includes the stimulation, collection and analysis of sweat. The standard of care sweat testing used at each institution will be compared to a new iontophoresis sweat test called the CF Quantum.

SUMMARY:
This is an observational comparative study to compare the standard-of-care methods for sweat testing used to support diagnosing cystic fibrosis (CF) against a new method of sweat testing called the CF Quantum Sweat Test System. The results of the new device in this study are for comparison ONLY and will NOT be used to diagnose, treat or mitigate the subject's condition.

DETAILED DESCRIPTION:
The primary objective is to evaluate the diagnostic accuracy of a new sweat test method in both normal individuals and individuals with CF or cystic fibrosis related metabolic syndrome (CRMS).

Subject participation is for one day and duration of study for each subject is one day. No follow-up will be required.

Number of subjects; 300 split evenly between subjects with previously diagnosed CF or CRMS (cystic fibrosis related metabolic syndrome) and subjects referred to the sweat test lab for clinical reasons.

Number of sites = 6, U of WI-Madison, U of WI-Milwaukee, U of MI-Ann Arbor, Dayton Children's Hospital (OH), U of MN, and Children's of Alabama.

Primary endpoints:

* Clinical and analytical sensitivity of the new test method
* Clinical and analytical sensitivity of the standard-of-care methods

Statistics Sensitivity and specificity will be calculated and reported along with the corresponding 95% confidence intervals. Bias assessment will be conducted according to the Clinical and Laboratory Standards Institute (CLSI) guidelines for method comparison and bias estimation. Pearson's correlation analysis will be conducted to test for adequate range of the replicate values for the new test method.

ELIGIBILITY:
Inclusion Criteria:

1. Patients referred to the sweat test lab on a clinical basis.
2. Infants who require a sweat test as follow-up to an abnormal CF screening test.
3. Patients who have already been diagnosed with CF or CRMS.
4. Written informed consent (and assent when applicable) obtained from subject or subject's legal representative.

Exclusion Criteria:

1. Patient is receiving oxygen by open delivery.
2. Infants less than 48 hours of age.
3. Diffuse inflammation or rash on the collection site.
4. Patients who have had a reaction to a prior iontophoretic sweat test procedure.
5. Arm is too small for both the new and conventional sweat test.

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: The study population includes those individuals with a previous diagnosis of CF or cystic fibrosis related metabolic syndrome (CRMS) and those individuals who have been referred to the sweat test lab for clinical reasons by a physician. The groups will be selected from the investigator's normal clinical practice.
Sampling Method: Probability Sample
Enrollment: 55 (Actual)
Dates: Start 2017-02-08 (Actual); Primary Completion 2018-07-01 (Actual); Study Completion 2018-07-01 (Actual)

PRIMARY OUTCOMES:
Diagnostic sensitivity and specificity (true positive rate and the false negative rate to measure chloride in the sweat sample) of the new sweat test device compared to the standard-of-care sweat test device | Day 1

SECONDARY OUTCOMES:
Compare the sweat test's "quantity not sufficient" (QNS) rate of the new device to the standard-of-care device. | Day 1

CONTACTS AND LOCATIONS:
Overall Officials: Michael Rock, MD, Principal Investigator — University of Wisconsin, Madison
Locations (6):
- United States (6):
  - Children's Hospital of Alabama at UAB, Birmingham, Alabama
  - Lurie Children's Hospital of Chicago, Chicago, Illinois
  - University of Michigan-Ann Arbor, Cystic Fibrosis Center, Ann Arbor, Michigan
  - University of Minnesota Masonic Children's Hospital, Minneapolis, Minnesota
  - Dayton Children's Hospital, Dayton, Ohio
  - University of Wisconsin-Madison CF Center, Madison, Wisconsin

IPD SHARING:
Plan to Share IPD: No